CLINICAL TRIAL: NCT00593866
Title: A Phase I/II Radiation Dose-Escalation Study of Intensity-Modulated Radiotherapy (IMRT) With Concurrent Gemcitabine in Patients With Unresectable Pancreatic Cancer
Brief Title: Dose-Escalation Study of Intensity-Modulated Radiotherapy(IMRT)in Patients With Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2006.018; IRB #HUM3315 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-08

CONDITIONS: Pancreatic Cancer
Keywords: Patients who have confirmed cancer arising from the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation Dose Escalation with Gemcitabine (Experimental): INTENSITY MODULATED RADIOTHERAPY
  Radiation dose escalation:
  Total dose Dose per fraction BED* Dose equivalent (1.8 Gy/fraction) Level 1 45.0 1.8 53.1 45.0 Level 2 50.0 2.0 60.0 50.4 Level 3 52.5 2.1 63.5 54.0 Level 4 55.0 2.2 67.1 57.0 Level 5 57.5 2.3 70.7 60.0 Level 6 60.0 2.4 74.4 63.0 Level 7 62.5 2.5 78.1 66.2 Level 8 65.0 2.6 81.9 69.4
  * BED=Biological Effective Dose; =10 Five fractions weekly, fraction size determined by dose level
  Gemcitabine:
  1000mg/m2 will be infused over 100 minutes on days 1, 8, 22 and 29 of the radiation treatment
  Interventions: Radiation: INTENSITY MODULATED RADIOTHERAPY; Drug: Gemcitabine

INTERVENTIONS:
Radiation: INTENSITY MODULATED RADIOTHERAPY — Five fractions weekly, fraction size determined by dose level
  Other Names: Radiation dose escalation:; Total dose Dose per fraction BED* Dose equivalent (1.8 Gy/fraction); Level 1 45.0 1.8 53.1 45.0; Level 2 50.0 2.0 60.0 50.4; Level 3 52.5 2.1 63.5 54.0; Level 4 55.0 2.2 67.1 57.0; Level 5 57.5 2.3 70.7 60.0; Level 6 60.0 2.4 74.4 63.0; Level 7 62.5 2.5 78.1 66.2; Level 8 65.0 2.6 81.9 69.4; * BED=Biological Effective Dose; =10
Drug: Gemcitabine — 1000mg/m2 will be infused over 100 minutes on days 1, 8, 22 and 29 of the radiation treatment

SUMMARY:
This is a research study for pancreatic cancer. One way of improving the results of current standard treatments is to try new approaches. This study will examine the use of a more advanced radiation therapy technique, called intensity modulated radiation therapy (IMRT), with chemotherapy. All subjects on this study will be treated with gemcitabine. This chemotherapy agent has been used for patients with pancreatic cancer. The researchers have already done studies using radiation therapy and gemcitabine. They want to build on the information they have from this previous research. The researchers want to find the best dose of IMRT that can be given at the same time that patients are receiving gemcitabine. To do this, they will vary the total dose of radiation received by patients on this study based on the information they have available from previously treated patients. The goal of the research is to identify the highest dose of IMRT that can be given at the same time as the chemotherapy without causing severe side effects.

ELIGIBILITY:
Inclusion Criteria:

* Is the patient 18 years of age or older.
* Does the patient have histologically or cytologically proven carcinoma of the pancreas
* Is the tumor unresectable or medically inoperable
* Does the patient have a Zubrod performance status of ≤ 2 (appendix I).
* Does the patient have an absolute neutrophil count of ≥ 1500/mm3, and platelets ≥ 100,000/mm3
* Does the patient have adequate renal function (creatinine < 2 mg/dl) and hepatic function (bilirubin < 3 mg/dl), with relief of biliary obstruction if present
* Is the patient free of significant co-morbid conditions that would preclude safe administration or completion of protocol therapy
* If the patient is of reproductive potential, has he or she agreed to use an effective method of contraception during treatment on this trial and for 6 months after treatment
* Is the patient aware of the investigational nature of the therapy such that they can provide written informed consent

Exclusion Criteria:

* Does the patient have a neuroendocrine tumor of the pancreas
* Does the patient have metastatic disease
* Does the patient have a history of abdominal radiation therapy
* Is there history of more than 1 month of therapy with single agent gemcitabine
* Has the patient used any investigational agent in the month before enrollment into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-06; Primary Completion 2012-05 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Zalupski, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - University Of Michigan, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Dose Escalation With Gemcitabine
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Dose Escalation With Gemcitabine
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 63 [48 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 40
  More than one race | 0
  Unknown or Not Reported | 4
Tumor Location [Number; unit: participants] — Location of tumor within the pancreas
  participants
    Head | 33
    Neck | 10
    Body/Tail | 7
Tumor Size [Median (Full Range); unit: centimeters (cm)] | 3.25 [1.6 to 7.1]
Tumor Volume [Median (Full Range); unit: Cubic Centimeter (cc)] | 47.9 [17 to 170]
Baseline CA 19-9 [Median (Full Range); unit: Units Per Millilitre (U/mL)] — The CA 19-9 is a simple blood test that measures the level of antigens in the blood serum of a person with pancreatic cancer.
  Units Per Millilitre (U/mL) | 102 [11 to 5028]

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Radiation Dose
Description: The maximum tolerated radiation dose delivered with intensity-modulated radiotherapy (IMRT) and concurrent gemcitabine in patients with unresectable adenocarcinoma of the pancreas.
Time Frame: 13 weeks post radiation
Measure: Number; unit: Gray (Gy)
Arm/Group | Radiation Dose Escalation With Gemcitabine
Number analyzed (Participants) | 50
Gray (Gy) | 55

2. Secondary Outcome: The Percentage of Participants Free From Local Progression at 2 Years
Time Frame: 2 Years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Dose Escalation With Gemcitabine
Number analyzed (Participants) | 50
percentage of participants | 59 [32 to 79]

ADVERSE EVENTS:
Arm/Group | Radiation Dose Escalation With Gemcitabine
Serious Adverse Events (participants affected / at risk) | 34/50
Other Adverse Events (participants affected / at risk) | 31/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Dose Escalation With Gemcitabine (N=50)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 8 (19)
Lymphopenia (Blood and lymphatic system disorders) | 11 (26)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 7 (18)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 6 (6)
Rigors/chills (General disorders) | 2 (2)
Weight loss (General disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (3)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Obstruction, GI, Stomach (Gastrointestinal disorders) | 1 (1)
Ulcer, GI, Duodenum (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hemorrhage, GI, Abdomen NOS (Vascular disorders) | 3 (4)
Hemorrhage, GI, Duodenum (Vascular disorders) | 1 (1)
Hemorrhage, GI, Varices (Vascular disorders) | 1 (2)
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 4 (5)
Liver dysfunction/failure (Hepatobiliary disorders) | 1 (1)
Infection with Grade 3 or 4 neutrophils, Abdomen (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophil, Blood (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils, Duodenum (Infections and infestations) | 1 (1)
Infection with Grade 3 or 4 neutrophils, Lung (Infections and infestations) | 1 (1)
Infection, Duodenum (Infections and infestations) | 1 (1)
Infection, Skin (Infections and infestations) | 2 (2)
Infection, Urinary Tract (Infections and infestations) | 1 (2)
Infection, Blood (Infections and infestations) | 1 (1)
Edema: limb (General disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (2)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3 (3)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (6)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Neurology - Other (Nervous system disorders) | 1 (1)
Pain, Abdomen (Gastrointestinal disorders) | 2 (2)
Pain, Chest (Cardiac disorders) | 1 (1)
Pain, Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Penis (Renal and urinary disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Dose Escalation With Gemcitabine (N=50)
Anemia (Blood and lymphatic system disorders) | 6 (15)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 22 (44)
Lymphopenia (Blood and lymphatic system disorders) | 24 (43)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 23 (45)
Platelets (Blood and lymphatic system disorders) | 6 (9)
Fatigue (General disorders) | 4 (5)
Fever (General disorders) | 6 (6)
Anorexia (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 5 (5)
Hemorrhage, GI (Vascular disorders) | 4 (5)
Hepatobiliary/Pancreas (Hepatobiliary disorders) | 6 (9)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 5 (6)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 5 (6)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 8 (11)
Pain, Abdomen (Gastrointestinal disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes